CLINICAL TRIAL: NCT02419924
Title: Proof of Concept: A Commode Assist Device for Excessive Perineal Descent
Brief Title: Proof of Concept: "Bottom's Up" Seat to Treat Constipation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-009864
Record Dates: First submitted 2015-04-06; First posted 2015-04-17 (Estimated); Results first posted 2020-09-02 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Constipation Aggravated; Pelvic Floor; Incompetency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental (Experimental): Pelvic floor support device to treat refractory constipation.
  Interventions: Device: "the Bottom's Up"

INTERVENTIONS:
Device: "the Bottom's Up" — A modified toilet seat that supports the perineum, preventing excessive pelvic floor descent and laxity which can cause constipation.
  Other Names: Pelvic floor support device to treat refractory constipation

SUMMARY:
Supporting the pelvic floor can reduce symptoms of constipation in patients with refractory constipation due to pelvic floor laxity and excessive perineal descent by means of a modified toilet seat, known as "the Bottom's Up".

DETAILED DESCRIPTION:
Efficacy and safety of a unique pelvic floor support device that fits into the Radiology defecography commode will be tested. Patients with refractory constipation due to known pelvic floor laxity and/or excessive perineal descent will be examined without, then with the device in place. Patients will complete questionnaires pertaining to device safety and efficacy before and after using the device. Radiographic images to document efficacy of support plus adequate emptying will be acquired during the study resulting in very low dose radiation exposure.

ELIGIBILITY:
10 Males and female subjects greater that 18 years of age with aggravated constipation due to pelvic floor laxity of at least 4 cm and excessive perineal descent of at least 4 cm will be evaluated.

Patients with constipation but no excessive laxity or descent will not be evaluated. Patients must be willing to sign consent, undergo defecography with and without "The Bottom's Up" device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-04; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Foxx-Orenstein, DO, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Experimental
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (18.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: The number of participants to report adverse events.
Time Frame: through study completion, approximately one day
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental
Number analyzed (Participants) | 12
Participants | 0

2. Secondary Outcome: Sense of Staining
Description: Sense of straining was measured using the self-reported answer to the modified Pelvic Floor Distress Inventory Questionnaire-20 (PFDI-20) question of 'Did you need to strain hard to empty your rectum'. The Likert scale questionnaire scores ranged from 0-10 where 0 = No, not at all and 10 = Yes, quite a bit.
Time Frame: post-defecography test, approximately 1 day
Population: Two subjects did not complete the questionnaire
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental
Number analyzed (Participants) | 10
score on a scale | 6.1 (2.8)

3. Secondary Outcome: Ease of Evacuation
Description: Ease of evacuation was measured using the self-reported answer to the modified Pelvic Floor Distress Inventory Questionnaire-20 (PFDI-20) question of 'Did you experience pain/discomfort when you emptied your rectum'. The Likert scale questionnaire scores ranged from 0-10 where 0 = No, not at all and 10 = Yes, quite a bit.
Time Frame: post-defecography test, approximately 1 day
Population: Two subjects did not complete the questionnaire
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental
Number analyzed (Participants) | 10
score on a scale | 2.9 (3.4)

4. Secondary Outcome: Completeness of Evacuation
Description: Completeness of evacuation was measured using the self-reported answer to the modified Pelvic Floor Distress Inventory Questionnaire-20 (PFDI-20) question of 'Did you feel that you completely emptied your rectum during this test'. The Likert scale questionnaire scores ranged from 0-10 where 0 = No, not at all and 10 = Yes, quite a bit.
Time Frame: post-defecography test, approximately 1 day
Population: Two subjects did not complete the questionnaire
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental
Number analyzed (Participants) | 10
score on a scale | 5.3 (3.0)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for the duration each subject was enrolled in the study, one day.
Arm/Group | Experimental
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-01): https://cdn.clinicaltrials.gov/large-docs/24/NCT02419924/Prot_SAP_000.pdf